CLINICAL TRIAL: NCT05891756
Title: Mesenteric Bacterial Translocation in Evolved Crohn's Disease
Acronym: MESENCROHN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Mutua de Terrassa (Other)
Responsible Party: Sponsor
Other Study IDs: MESENCROHN
Record Dates: First submitted 2023-05-11; First posted 2023-06-07 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Crohn Disease
Keywords: Crohn Disease; Mesenteric fat; Bacterial translocation; Innate immunity; Genetic polymorphisms
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Mesenteric fat, ileal tissue and whole blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CD patients requiring surgical treatment (ileocecal resection)
- Control group: Patients requiring an ileocecal resection for a cause other than CD

SUMMARY:
Mesenteric fat can be invaded by gut bacteria through a process called bacterial translocation, which is the invasion of viable bacteria from the gastrointestinal tract to extraintestinal sites (mesenteric lymph nodes, liver, spleen, kidney, bloodstream, etc.). In Crohn's disease (CD), bacterial translocation could increase the disproportionate inflammatory response already present and contribute to disease progression by stimulating the production of pro-inflammatory cytokines and immune-cell infiltration in the mesentery. Several mechanisms may promote bacterial translocation, such as bacterial overgrowth, disruption of the intestinal mucosal barrier and alterations in the immune system.

Ileocecal surgical resection is required in some patients with complicated or refractory CD. Unfortunately, post-surgical disease recurrence happens in up to 40% of cases, probably defining a subgroup of CD patients with a particular aggressive form of the disease. The complete microbiome (in gastrointestinal and extraintestinal sites) in CD patients that develop early post-surgical recurrence, as well as the association to innate immunity alterations, has not yet been studied.

The primary aim of the study is to explore the bacterial microbiome of CD patients and its association with early post-surgical recurrence and clinical or genetic variables related to innate immunity. To achieve this, the bacterial DNA present in mesenteric fat and ileal tissue (inflamed and non-inflamed) from surgical resection samples as well as blood samples from CD patients will be studied. Genetic polymorphisms, relevant clinical data and disease recurrence will also be evaluated.

The investigators hypothesize that bacterial translocation to the mesentery fat near the inflamed intestine is one of the mechanisms for perpetuation and chronicity of inflammation and therefore post-surgical recurrence in CD. The investigators expect to find a distinctive bacterial profile (in quantity and quality) in the mesenteric fat of patients with early post-surgical recurrence and/or with genetic variants that cause alterations in innate immunity.

The study of the microbiome in CD could help to identify the patients with a more aggressive disease form that will probably present early post-surgical recurrence, and could raise the possibility of microbial modulation as therapy for CD.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 years or older)
* Informed consent signed
* To require an ileocecal resection as part of the treatment of Crohn's Disease
* In the case of controls: not having Inflammatory Bowel Disease and requiring an ileocecal resection for another reason

Exclusion Criteria:

* To require an ileocecal resection with definitive or transient ileostomy
* In the case of controls: existence of a family history of Inflammatory Bowel Disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from the Hospital Universitari MútuaTerrassa
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Differences in the proportions and abundance of bacterial taxa (defined as total percentage of bacterial DNA sequences) between the mesentery, ileal tissue and blood between CD patients with and without early post-surgical disease recurrence | at inclusion (surgery)
Differences in the function of the bacterial profile (defined as the metagenome function analysis) between the mesentery, ileal tissue and blood between CD patients with and without early post-surgical disease recurrence | at inclusion (surgery)

SECONDARY OUTCOMES:
Association analysis of genetic variants related to innate immunity and the bacterial microbiome profile of CD patients | at inclusion (surgery)
  DNA polymorphisms detection in blood: ATG16L1 (rs2241880, rs3792109, rs3828309); NOD2 / CARD15 (rs2066844, rs2066845) and IRGM (rs13361189, rs4958847, rs1336119, rs10065172, rs7714584).

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitari MútuaTerrassa, Terrassa, Barcelona, Spain

REFERENCES:
- [Background] Schaffler A, Scholmerich J. Innate immunity and adipose tissue biology. Trends Immunol. 2010 Jun;31(6):228-35. doi: 10.1016/j.it.2010.03.001. PMID 20434953
- [Background] Batra A, Heimesaat MM, Bereswill S, Fischer A, Glauben R, Kunkel D, Scheffold A, Erben U, Kuhl A, Loddenkemper C, Lehr HA, Schumann M, Schulzke JD, Zeitz M, Siegmund B. Mesenteric fat - control site for bacterial translocation in colitis? Mucosal Immunol. 2012 Sep;5(5):580-91. doi: 10.1038/mi.2012.33. Epub 2012 May 9. PMID 22569302
- [Background] Bertin B, Desreumaux P, Dubuquoy L. Obesity, visceral fat and Crohn's disease. Curr Opin Clin Nutr Metab Care. 2010 Sep;13(5):574-80. doi: 10.1097/MCO.0b013e32833cf0f4. PMID 20625283
- [Background] Alexander JW, Boyce ST, Babcock GF, Gianotti L, Peck MD, Dunn DL, Pyles T, Childress CP, Ash SK. The process of microbial translocation. Ann Surg. 1990 Oct;212(4):496-510; discussion 511-2. doi: 10.1097/00000658-199010000-00012. PMID 2222015
- [Background] Laffineur G, Lescut D, Vincent P, Quandalle P, Wurtz A, Colombel JF. [Bacterial translocation in Crohn disease]. Gastroenterol Clin Biol. 1992;16(10):777-81. French. PMID 1478405
- [Background] Zulian A, Cancello R, Micheletto G, Gentilini D, Gilardini L, Danelli P, Invitti C. Visceral adipocytes: old actors in obesity and new protagonists in Crohn's disease? Gut. 2012 Jan;61(1):86-94. doi: 10.1136/gutjnl-2011-300391. Epub 2011 Sep 19. PMID 21930728
- [Background] Shi H, Kokoeva MV, Inouye K, Tzameli I, Yin H, Flier JS. TLR4 links innate immunity and fatty acid-induced insulin resistance. J Clin Invest. 2006 Nov;116(11):3015-25. doi: 10.1172/JCI28898. Epub 2006 Oct 19. PMID 17053832
- [Background] Siegmund B. Mesenteric fat in Crohn's disease: the hot spot of inflammation? Gut. 2012 Jan;61(1):3-5. doi: 10.1136/gutjnl-2011-301354. Epub 2011 Nov 7. No abstract available. PMID 22068165
- [Background] Sokol H, Brot L, Stefanescu C, Auzolle C, Barnich N, Buisson A, Fumery M, Pariente B, Le Bourhis L, Treton X, Nancey S, Allez M, Seksik P; REMIND Study Group Investigators. Prominence of ileal mucosa-associated microbiota to predict postoperative endoscopic recurrence in Crohn's disease. Gut. 2020 Mar;69(3):462-472. doi: 10.1136/gutjnl-2019-318719. Epub 2019 May 29. PMID 31142586
- [Background] Domenech E, Manosa M, Bernal I, Garcia-Planella E, Cabre E, Pinol M, Lorenzo-Zuniga V, Boix J, Gassull MA. Impact of azathioprine on the prevention of postoperative Crohn's disease recurrence: results of a prospective, observational, long-term follow-up study. Inflamm Bowel Dis. 2008 Apr;14(4):508-13. doi: 10.1002/ibd.20359. PMID 18183602
- [Background] Gutierrez A, Scharl M, Sempere L, Holler E, Zapater P, Almenta I, Gonzalez-Navajas JM, Such J, Wiest R, Rogler G, Frances R. Genetic susceptibility to increased bacterial translocation influences the response to biological therapy in patients with Crohn's disease. Gut. 2014 Feb;63(2):272-80. doi: 10.1136/gutjnl-2012-303557. Epub 2013 Feb 1. PMID 23376290
- [Background] Li Y, Zuo L, Zhu W, Gong J, Zhang W, Gu L, Guo Z, Li N, Li J. The impact of bacterial DNA translocation on early postoperative outcomes in Crohn's patients undergoing abdominal surgery. J Crohns Colitis. 2015 Mar;9(3):259-65. doi: 10.1093/ecco-jcc/jju029. Epub 2015 Jan 2. PMID 25555386
- [Background] Takesue Y, Ohge H, Uemura K, Imamura Y, Murakami Y, Yokoyama T, Kakehashi M, Sueda T. Bacterial translocation in patients with Crohn's disease undergoing surgery. Dis Colon Rectum. 2002 Dec;45(12):1665-71. doi: 10.1007/s10350-004-7256-z. PMID 12473892
- [Background] Kosovac K, Brenmoehl J, Holler E, Falk W, Schoelmerich J, Hausmann M, Rogler G. Association of the NOD2 genotype with bacterial translocation via altered cell-cell contacts in Crohn's disease patients. Inflamm Bowel Dis. 2010 Aug;16(8):1311-21. doi: 10.1002/ibd.21223. PMID 20232407
- [Background] Kiernan MG, Coffey JC, McDermott K, Cotter PD, Cabrera-Rubio R, Kiely PA, Dunne CP. The Human Mesenteric Lymph Node Microbiome Differentiates Between Crohn's Disease and Ulcerative Colitis. J Crohns Colitis. 2019 Jan 1;13(1):58-66. doi: 10.1093/ecco-jcc/jjy136. PMID 30239655